CLINICAL TRIAL: NCT01907880
Title: A Randomized, Double-blind, Placebo-controlled, Phase IV Trial Evaluating the Palliative Benefit of Either Continuing Pamidronate or Switching to Second-line Zoledronic Acid in Breast Cancer Patients With High-risk Bone Metastases.
Brief Title: The ODYSSEY TRIAL Phase IV Trial Evaluating the Palliative Benefit of Pamidronate or Zoledronic Acid in Breast Cancer
Acronym: ER11-03
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: Canadian Breast Cancer Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2011349-01H
Record Dates: First submitted 2013-07-22; First posted 2013-07-25 (Estimated); Last update posted 2017-07-07 (Actual); Status verified 2016-09

CONDITIONS: Breast Cancer
Keywords: breast; bone; pain
MeSH Terms: conditions — Breast Neoplasms; Pain | interventions — Pamidronate; Zoledronic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pamidronate and placebo (Active Comparator): Patients will receive two infusions simultaneously, at each study visit, one of Pamidronate and another of the placebo. After completing 3 cycles of study treatment, patients will resume their monthly intravenous pamidronate infusions as per current standard of care.
  Interventions: Drug: Pamidronate; Drug: placebo
- Zoledronic acid and placebo (Active Comparator): Patients will receive two infusions simultaneously, at each study visit, one of Zoledronic acid and another of the placebo. After completing 3 cycles of study treatment, patients will resume their monthly intravenous pamidronate infusions as per current standard of care.
  Interventions: Drug: Zoledronic acid; Drug: placebo

INTERVENTIONS:
Drug: Pamidronate — 90mg IV once every 4 weeks for 3 cycles
  Other Names: ADP Sodium; Aredia®
  Arms: Pamidronate and placebo
Drug: Zoledronic acid — 4mg IV every 4 weeks for 3 cycles
  Other Names: Reclast; Zometa; Aclasta
  Arms: Zoledronic acid and placebo
Drug: placebo

SUMMARY:
Metastatic breast cancer patients with bone involvement who are at high-risk of subsequent skeletal related event (SRE), defined as radiotherapy or surgery to the bone, pathological fracture, spinal cord compression, or hypercalcemia (as reflected through: elevated sCTX or bone pain or a prior SRE despite receiving standard bisphosphonate therapy) should experience a decrease in the surrogate marker, sCTX, at week 12 if switched to zoledronic acid compared with those patients who continue on intravenous pamidronate (i.e. current standard of care). The investigators propose that a drop in sCTX will correlate with improved pain, quality of life and a reduced incidence of further SREs.

DETAILED DESCRIPTION:
This study will be a prospective, randomized, double-blind, placebo controlled, Phase IV study of pamidronate vs. zoledronic acid in women with breast cancer and bone metastases. Patients who are at high-risk of subsequent SREs will be screened for entry into this study. High-risk will be defined as fulfilling one or more of the following criteria: elevated sCTX (>400ng/L) and/or bone pain and/or a prior SRE and/or progression of bone disease (by imaging) despite at least 3 months of pamidronate therapy. Patients who meet the eligibility criteria, will be randomized to receive 3 cycles of intravenous zoledronic acid (4mg intravenously over 15 minutes) or to continue their standard dose of pamidronate. Both treatments will be given at 4 week intervals. Patients will be stratified according to whether or not they have had a SRE prior to study entry, progressive bone disease or bone pain. In order for the study to be double-blind, patients will receive two infusions simultaneously, at each study visit, one of the active drug and another of the placebo. After completing 3 cycles of study treatment, patients will resume their monthly intravenous pamidronate infusions as per current standard of care.

ELIGIBILITY:
Inclusion Criteria:

1. Metastatic breast cancer to the bone with radiologically confirmed bone metastases
2. High-risk of subsequent SRE as reflected through either: elevated serum CTX (> 400ng/L) and/or bone pain (using BPI) and/or prior SRE while on bisphosphonate therapy and/or progressive bone metastasis (by imaging)
3. On pamidronate therapy for at least 3 months
4. ECOG ≤ 2 and life expectancy > 3 months
5. Serum creatinine ≤ 2.0 × ULN (zoledronic acid or pamidronate to be renal dosed as per institution standard)
6. No changes in systemic treatment in the 4 weeks prior to study entry or anticipated changes in the 4 weeks after entering the study. Markers of bone formation can be affected by a change in systemic therapies
7. Ability to take calcium and Vitamin D as per Health Canada recommended daily doses for the duration of the study
8. Ability to provide informed consent and complete study evaluations.

Exclusion Criteria:

1. Patients with acute symptomatic pathological fractures or acute spinal cord compression until such time as the appropriate management (surgery and/or radiotherapy) has been completed
2. Acute hypercalcemia (>3.5 mmol/L)
3. Hypersensitivity to any bisphosphonate
4. Patients with rapidly progressive non-bone metastases for whom delaying a change in systemic anti-cancer treatment for the 1 month biochemical marker evaluation period could have a detrimental impact on patient outcome.
5. Renal dysfunction (≥ 2x creatinine of the upper limit of normal )
6. Pregnancy or lactation
7. Patients with dental abscesses or patients potentially requiring tooth extraction while on study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2012-08; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
sCTX values | baseline, 1 week post treatment, week 4, week 8, week 12
  To compare the proportion of high-risk metastatic breast cancer patients with bone metastases that will achieve a decrease in sCTX (surrogate for decrease risk of SREs) in the zoledronic and pamidronate treatment arms.

SECONDARY OUTCOMES:
Palliative response | baseline, week 1, week 4, week 8, week 12.
  To determine the proportion of high-risk metastatic breast cancer patients that will achieve a significant improvement in palliative response (18) (defined as a two unit drop in their worst pain score, based on a brief pain inventory questionnaire for two consecutive measurements at least one month apart) in the zoledronic and pamidronate treatment arms.

OTHER OUTCOMES:
predictor of pain benefit | week 1 and week 12
  To assess whether a drop in sCTX one week post infusion of zoledronic acid is a predictor of pain benefit at week 12. We will test the strength of the association in sCTX drop (any drop from baseline level) at week 1 and palliative response when measured at week 12, using the validated BPI and FACT-BP questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Mark Clemons, Dr., Principal Investigator — The Ottawa Hospital
Locations (1):
- The Ottawa Hospital Cancer Centre, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
results will be published.